CLINICAL TRIAL: NCT06021886
Title: CS Scar Impact on ART Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: HealthPlus Fertility Center (Other)
Responsible Party: Principal Investigator, Ahmed Elsayed Hassan Hamed Elbohoty, Reproductive medicine consultant, HealthPlus Fertility Center
Other Study IDs: REC/2023/P38
Record Dates: First submitted 2023-06-21; First posted 2023-09-01 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Fertility Issues
Keywords: CS Scar Impact on ART Outcomes
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patient without scar: history of euploid embryo transfer
- patient with cs scar no Niche: history of euploid embryo transfer
- patient with cs scar with niche: history of euploid embryo transfer

SUMMARY:
CS scar impact on ART outcomes, Retrospective Cohort Study IVF outcome can be affected by the presence of caesarean section scar with or without defect in different ways

DETAILED DESCRIPTION:
CS scar impact on ART outcomes, Retrospective Cohort Study IVF outcome can be affected by the presence of caesarean section scar with or without defect in different ways; increase difficulty of embryo transfer, presence intrauterine fluid at the time of transfer can affect the chances of embryo implantation and increase the rate of spontaneous miscarriages To compare the success rates and outcomes of pregnancies of frozen embryo transfer for euploid embryos in patients without caesarean section, and who had caesarean section (with or without a NICHE) after euploid embryo transfer. Does CS scar and CS scar defect affect IVF outcome? All women who underwent an embryo transfer with a Euploid embryo between 2015 and 2022, who meet the inclusion criteria will be included in the study.

* Inclusion Criteria: Age 25-40 years old. Euploid embryo transfer. Medically free BMI less tha 30 kg/m2 Hormone therapy preparation for FET.
* Exclusion criteria Previous uterine scar other than cesarean section. Congenital uterine abnormalities Presence of intrauterine lesions e.g., polyp, fibroid, Endometriosis or adenomyosis Hydrosalpinx, Chronic endometritis
* Primary outcome: Clinical pregnancy rate, defined as a pregnancy with a detectable heart rate at 7 weeks of gestation or beyond.
* Secondary outcomes : Early pregnancy complications Ectopic pregnancy or Miscarriage. Caesarean section scar dehiscence or

ELIGIBILITY:
Inclusion Criteria:

* Age 25-40 years old.

Euploid embryo transfer.

Medically free

BMI less tha 30 kg/m2

Hormone therapy preparation for FET.

Exclusion Criteria:

- Exclusion criteria

Previous uterine scar other than cesarean section.

Congenital uterine abnormalities

Presence of intrauterine lesions e.g., polyp, fibroid,

Endometriosis or adenomyosis

Hydrosalpinx, Chronic endometritis

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: All women who underwent an embryo transfer with a Euploid embryo between 2005 and 2022, who meet the inclusion criteria will be included in the study. To compare the success rates and outcomes of pregnancies of frozen embryo transfer for euploid embryos in patients without caesarean section, and who had caesarean section (with or without a NICHE) after euploid embryo transfer.
Sampling Method: Probability Sample
Enrollment: 510 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
CS scar impact on ART outcomes, Retrospective Cohort Study | 2015 to 2022,
  Clinical pregnancy rate

SECONDARY OUTCOMES:
ART outcomes | 2015 to 2022,
  Early pregnancy complications:
  Ectopic pregnancy or Miscarriage.
  Caesarean section scar dehiscence or rupture.
  Presence of intrauterine fluid accumulation at the time of ET.
  Endometrial thickness at the time of ET.
  Live birth.

CONTACTS AND LOCATIONS:
Locations (1):
- HealthPlus fertility Centre, Abu Dhabi, United Arab Emirates